CLINICAL TRIAL: NCT03413462
Title: Multi-center,Randomized,Double Blind,Placebo Controlled,Efficacy and Safety Study of HS-25 in Adults With Primary Hypercholesterolemia
Brief Title: Efficacy and Safety Study of HS-25 in Chinese Adults With Primary Hypercholesterolemia
Acronym: HS-25-III-01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-25-III-01
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-01

CONDITIONS: Primary Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-25 (Active Comparator): 20mg, QD, 12 weeks
  Interventions: Drug: HS-25
- Placebo of HS-25 (Placebo Comparator): 20mg, QD, 12 weeks
  Interventions: Drug: HS-25; Drug: Placebo of HS-25

INTERVENTIONS:
Drug: HS-25 — HS-25 10mg/tablet, 20mg,once daily,for 12 weeks, and then HS-25 20mg once daily for 40 weeks.
Drug: Placebo of HS-25 — Placebo HS-25 10mg/tablet, 20mg,once daily,for 12 weeks,and then HS-25 20mg once daily for 40 weeks.
  Arms: Placebo of HS-25

SUMMARY:
To determine the efficacy of HS-25 (20mg) in reducing low density lipoprotein-cholesterol (LDL-C) levels after a 12-week period of treatment in adults with primary hypercholesterolemia;

To determine the safety of HS-25 (20mg) in subjects with LDL-C

DETAILED DESCRIPTION:
This is a 12-week, randomized, double-blind, placebo-controlled study designed to assess the effects of the cholesterol absorption inhibitor HS-25 on LDL-C levels in adults who have untreated LDL-C levels ranging from 3.36-4.88mmol/L(130-189 mg/dL)and fasting triglyceride levels < 350 mg/dL. Eligibility is restricted to 18-75 years old men or women who are using a highly effective birth control method or are not of childbearing potential. Patients with diabetes, a history of myocardial infarction or other clinical evidence of atherosclerotic vascular disease are not eligible for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 18 to 75 years of age, male or female using a highly effective birth control method or not of child-bearing potential, at Visit 1 (screening visit).
* LDL-C 130 to 189 mg/dL (inclusive) on a cholesterol lowering diet but no lipid modifying drug treatment for at least 6 weeks.
* A qualifying LDL-C value must be obtained at the beginning and end of the placebo run-in (Visit 2 and Visit 3) and the Visit 3 value must be within 12% of the value at Visit 2, higher or lower; the average of both qualifying values must be in the range of 130 to 189 mg/dL (inclusive) for inclusion in the study.
* TG ≤ 350 mg/dL on a cholesterol lowering diet but no lipid modifying drug treatment for at least 6 weeks and TG levels must be ≤ 350 mg/dL at both Visit 2 and Visit 3
* Signed written informed consent.

Exclusion Criteria:

* Liver transaminases > 1.5 x upper limit of normal.
* Homozygous Familial Hypercholesterolemia.
* Subject who was diagnosed as diabetes with aged greater than 40 years old.
* Subject who was diagnosed as diabetes with one of the following of cardiovascular risk factorss: Hypertention Bp ≥ 140/90mmHg,or smoking, or low HDL-C (1.04mmol/L), or BMI≥28kg/m2.
* Women who are pregnant or breast feeding.
* Atherosclerotic cardiovascular disease including Arteriosclerotic heart disease, Acute coronary syndrome，Coronary artery bypass graft,Coronary angioplastyPeripheral arteriosclerosis,Cerebrovascular accident
* history of Severe Endiocrine disease (for example Thyroid function abnormal)
* History of a positive test for human immunodeficiency virus, hepatitis B or hepatitis C.
* History of advanced cancer
* Arrhythmias need to be treated by medications
* Had severe injured or surgery in 6 months before study start.
* Hypersensitive to HS-25 or place.
* History of intolerance to ezetimibe.
* Participation other studies in three months.
* Treatment with a fibric acid derivative (eg, fenofibrate, gemfibrozil), probucol, warfarin, systemic corticosteroid, cyclosporine or other immunosuppressant agent within the prior 12 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
LDL-C | 2,4,8,12,18,24,38,52 weeks
  Percent change from baseline in LDL-C after 2,4,8,12,18,24,38,52 weeks of double-blind treatment

SECONDARY OUTCOMES:
Non-HDL-C | 2,4,8,12,18,24,38,52 weeks
  Percent change from baseline in LDL-C after 2,4,8,12,18,24,38,52 weeks of double-blind treatment
HDL-C | 2,4,8,12,18,24,38,52 weeks
  Percent change from baseline in LDL-C after 2,4,8,12,18,24,38,52 weeks of double-blind treatment
TC | 2,4,8,12,18,24,38,52 weeks
  Percent change from baseline in LDL-C after 2,4,8,12,18,24,38,52 weeks of double-blind treatment
TG | 2,4,8,12,18,24,38,52 weeks
  Percent change from baseline in LDL-C after 2,4,8,12,18,24,38,52 weeks of double-blind treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, Principal Investigator — Peking University First Hospital